CLINICAL TRIAL: NCT04692987
Title: Effectiveness of Decision-aid Video on Colorectal Cancer Screening in Primary Healthcare Setting: A Randomized Controlled Trial
Brief Title: Effectiveness of Decision-aid Video on Colorectal Cancer Screening
Acronym: DAVOCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Azmawati, Public Health Specialist & Medical Lecturer, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: FF-2020-155
Record Dates: First submitted 2020-12-22; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Cancer
Keywords: Screening; Primary care; Video
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial will be conducted in 3 months duration, with intention-to-treat.
Who Masked: Participant, Care Provider
Masking Description: Investigators will designate participants to which arm using random sampling. Participants and care providers are masked to which arm they receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive decision-aid video
  Interventions: Other: Decision-aid video
- Usual care (No Intervention): Participants will receive usual care

INTERVENTIONS:
Other: Decision-aid video — Decision-aid video will be developed to disseminate knowledge and to raise awareness on colorectal cancer screening
  Arms: Intervention

SUMMARY:
Colorectal cancer (CRC) is the second most common cancer in Malaysia. Diagnosing CRC at early stage is crucial to reduce their mortality risk. To achieve this aim, CRC screening promotion intervention is deemed necessary.

DETAILED DESCRIPTION:
High-quality CRC screening interventions and approaches should be delivered to a large proportion of target population.

To our knowledge, there is no interactive video been developed, that can be used as educational tool for CRC screening in Malaysia. By developing an educational video, we hope that it can be used by health professionals to promote CRC screening, favoring their empowerment for prevention and control of disease.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian aged 50 - 74 years old
* No previous history or family history of CRC
* Asymptomatic of CRC
* Never participated in CRC screening

Exclusion Criteria:

* Acute patients
* Patients on aspirin, warfarin or any blood-thinning agent
* Illiterate or having a significant vision or hearing impairment

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with colorectal cancer screening completion | 3 months
  Number of participants with completion of fecal occult blood test or colonoscopy procedures by participants

SECONDARY OUTCOMES:
Number of participants with colonoscopy completion among those with positive fecal occult blood test | 3 months
  Number of participants who are completed colonoscopy among those positive fecal occult blood test
Period time from intervention to fecal occult blood test uptake | 3 months
  Duration taken after received intervention to screening uptake
Barriers towards the colorectal cancer screening uptake | 3 months
  List of barriers (numbers) towards the colorectal cancer screening uptake

CONTACTS AND LOCATIONS:
Overall Officials: Azmawati Mohammed Nawi, Principal Investigator — The National University of Malaysia
Locations (1):
- The National University of Malaysia, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
Only three principal investigators will have access to participants' data